CLINICAL TRIAL: NCT04987918
Title: Gazelle COVID-19 Test Clinical Accuracy Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hemex Health (Industry)
Responsible Party: Sponsor
Other Study IDs: GZL-FC10-PTL-0001
Record Dates: First submitted 2021-07-30; First posted 2021-08-03 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Applied Biosystems TaqPath COVID- 19 Combo Kit — Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)

SUMMARY:
Gazelle COVID-19 is a fluorescent lateral flow immunoassay and accompanying Reader intended for the qualitative detection of nucleocapsid antigen from SARS-CoV-2 in nasal swab specimens from individuals who are suspected of COVID-19 by their healthcare provider within 5 days of symptom onset. The study will be conducted To obtain data to measure the positive percent agreement and negative percent agreement of the Gazelle COVID-19 Test compared to Reverse Transcriptase Polymerase Chain Reaction (RT-PCR).The study will assess Gazelle COVID-19 Test performance using dual mid-turbinate nasal swab samples. This study will primarily assess Gazelle COVID-19 Test performance on symptomatic subjects (within five days of onset of symptoms) at point of care (POC). A subset of asymptomatic subjects will be enrolled after the symptomatic subject enrollment is complete.

ELIGIBILITY:
Symptomatic study:

Inclusion Criteria:

The presence of clinical signs and symptoms consistent with COVID-19. Signs and symptoms include:

* Fever
* Coughing
* Shortness of breath
* Recent loss of sense of smell or taste
* Chills
* Repeated shaking with chills
* Muscle pain
* Headache
* Sore throat
* Vomiting or diarrhea

  * Within 1-5 days of symptom onset
  * Informed consent for all the samples will be obtained from the subject or obtained from the parent/guardian in case the patient is a minor
  * All ages
  * All genders
  * Pregnant women

Exclusion Criteria:

* Severe disease requiring immediate medical intervention
* Inability to tolerate sampling procedure (nasal swab)
* Failure to provide informed consent
* Nasal deformities preventing sampling by swab
* Ongoing nosebleeds or use of a nasal spray within the last 4 hours.
* Asymptomatic patients

Asymptomatic study:

Inclusion criteria:

* Present to the facility for a COVID-19 test without symptoms
* Informed consent for all specimens will be obtained from the patient or obtained from the parent/guardian in case the patient is a minor

Exclusion Criteria:

Exclusion criteria include one or more of the following:

* Severe disease requiring immediate medical intervention
* Inability to tolerate sampling procedure
* Is below 2 years old
* Failure to provide informed consent
* Nasal deformities preventing sampling by swab
* Ongoing nosebleeds or use of a nasal spray within the last 4 hours.
* Presence of typical symptoms of COVID-19 (fever, sore throat, fatigue, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive subjects of all ages who visit the facility for covid 19 testing (symptomatic and asymptomatic).
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Positive percent agreement and negative percent agreement of the Gazelle COVID-19 Test compared to Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) will be measured | 3 months

SECONDARY OUTCOMES:
Sensitivity and specificity on at least 30, maximum 65, SARS-CoV-2 positive patient samples will be assessed | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Robert Fortna, MD, PhD, Principal Investigator — Northwest Pathology
Locations (1):
- Northwest Pathology drive thru site, Bellingham International Airport, Bellingham, Washington, United States